CLINICAL TRIAL: NCT04722237
Title: Acceptance and Commitment Therapy for Young Brain Tumour Survivors: An Acceptability and Feasibility Trial
Brief Title: Acceptance and Commitment Therapy for Neuro-Oncology Wellbeing
Acronym: ACT NOW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Nottingham (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); University of Exeter (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University of Surrey (Other); Newcastle University (Other); University of Bristol (Other); DNA-v International (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 266746
Record Dates: First submitted 2020-11-26; First posted 2021-01-25 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Brain Tumors; Quality of Life; Brain Tumor, Pediatric
Keywords: Acceptance and Commitment Therapy; Cancer; Oncology; Quality of survival; children and adolescents
MeSH Terms: conditions — Brain Neoplasms; Neoplasms | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: This study is a two-arm, parallel group, randomised controlled trial comparing ACT with waitlist controls who will then receive ACT after the 3-month waiting period. Participants will be randomised on a 1:1 ratio to receive 12-weeks of treatment either immediately or following a 12-week wait. The treatment will be DNA-v which is a model of ACT adapted to those aged 11-24 years. The model will be further adapted for those who have undergone brain tumour treatment. As trial therapists will perform assessments, blinding is not possible. Follow-up assessments will be conducted at 12-, 24-, 36-, and 48-weeks post-randomisation with primary end point at 12-weeks.
Masking Description: As trial therapists will perform assessments, blinding is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Acceptance and Commitment Therapy (Experimental): Receiving 6-to-12 weekly sessions of Acceptance and Commitment Therapy immediately after allocation. Each session will be up to one hour in length.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Waitlist Control (No Intervention): Receiving no intervention during a 12-week wait, though no restrictions will be placed on the use of other services. After the wait participants will receive 6-to-12 weekly sessions of Acceptance and Commitment Therapy. Each session will be up to one hour in length.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy (ACT) is an evidence-based psychological therapy that has been used to improve physical and mental health among adults with health conditions, including cancer (Graham, Gouick, Krahe, & Gillanders, 2016). It fosters engagement with, rather than avoidance of, painful experiences, to move towards acceptance of unchangeable difficulties alongside building a rich and meaningful life despite the presence of ongoing problems.
  Arms: Immediate Acceptance and Commitment Therapy

SUMMARY:
Background. Survivors of childhood brain tumours have the poorest health-related quality of life of all cancer survivors due to the multiple physical and psychological sequelae of brain tumours and their treatment. Remotely delivered Acceptance and Commitment Therapy (ACT) may be a suitable and accessible psychological intervention to support young people who have survived brain tumours.

Aims. This study aims to assess the feasibility and acceptability of remotely delivered ACT to improve quality of life among young brain tumour survivors.

Method. This study is a two-arm, parallel group, randomised controlled trial comparing ACT with waitlist control. Participants will be aged 11-24 years and survivors of brain tumours who have completed cancer treatment. Participants will be randomised to receive 12 weeks of ACT either immediately or after a 12-week wait. The durability of treatment effects will be assessed by further follow-up assessments at 24-, 36- and 48- weeks. The DNA-v model of ACT will be employed, which is a developmentally appropriate model for young people. Feasibility will be assessed using the proportion of those showing interest who consent to the trial and complete the intervention. A range of clinical outcome measures will also assess physical and mental health, everyday functioning, quality of life and service usage. Acceptability will be assessed using participant evaluations of the intervention, alongside qualitative interviews and treatment diaries analysed thematically.

Discussion. This study will provide an initial assessment of the value of remotely delivered ACT in supporting recovery and coping for young people after brain tumour treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 11-to-24 years at the time of randomisation
* Received treatment for a brain tumour at a participating Principle Treatment Centre
* Active brain tumour treatment is complete and their condition stable for at least six-months
* Have sufficient cognitive ability to engage with ACT sessions as judged by the clinician at baseline assessment
* competent to provide informed consent (participants aged 16 or over) or assent (participants aged 11-15)
* Parent/carer competent to provide informed consent (for participants aged 11-15)

Exclusion Criteria:

* Received a structured behavioural intervention within six-months prior to study recruitment
* Previous or current alcohol/substance dependence, psychosis, suicidality, or eating disorder
* Moderate or severe intellectual disability, confirmed through researcher judgement at screening through questions relating to school type and previous diagnoses
* Immediate risk to self or others
* The patient or their parent/carer is not able to speak, read or write English

Ages: 11 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Treatment completion rate | assessed at 3-month follow-up
  The proportion of patients showing interest who then consent to the trial and complete the intervention
Treatment completion rate | assessed at 6-month follow-up
  The proportion of patients showing interest who then consent to the trial and complete the intervention
Session attendance rate | assessed at 3-month follow-up
  The session attendance rate compared to feasibility benchmarks
Session attendance rate | assessed at 6-month follow-up
  The session attendance rate compared to feasibility benchmarks
The credibility/expectancy questionnaire | Assessed at baseline
  Assessing participant ratings of treatment credibility. Minimum score = 5; maximum score = 45. Higher scores indicate better outcome.
The credibility/expectancy questionnaire | Assessed at session 2
  Assessing participant ratings of treatment credibility. Minimum score = 5; maximum score = 45. Higher scores indicate better outcome.
The experience of service questionnaire | Assessed at 3-month follow-up.
  A questionnaire used nationally in child and adolescent mental health services completed by patients and parents/carers (if under 16) to assess participants' experience of the intervention. An additional item has been added to the experience of service questionnaire to assess video-conferencing treatment satisfaction. Minimum score = 0; maximum score = 20. Higher scores indicate better outcome.
The experience of service questionnaire | Assessed at 6-month follow-up.
  A questionnaire used nationally in child and adolescent mental health services completed by patients and parents/carers (if under 16) to assess participants' experience of the intervention. An additional item has been added to the experience of service questionnaire to assess video-conferencing treatment satisfaction. Minimum score = 0; maximum score = 20. Higher scores indicate better outcome.

SECONDARY OUTCOMES:
Acceptance and Action Questionnaire II | assessed at 3, 6, 9 and 12-month follow-up
  A brief 7-item self-report measure assessing psychological inflexibility, which is the central treatment target for ACT. Validated for use among patients aged 16 and over. Minimum score = 7; maximum score = 49. Higher scores indicate worse outcome.
Avoidance and Fusion Questionnaire for Youth 8-items | assessed at 3, 6, 9 and 12-month follow-up
  A brief self-report measure of psychological inflexibility, for children (11 to 15 year old participants). Minimum score = 0; maximum score = 32. Higher scores indicate worse outcome.
World Health Organisation wellbeing index 5-items | assessed at 3, 6, 9 and 12-month follow-up
  A brief self-reported assessment of wellbeing and mental health. Minimum score = 7 score; maximum = 49. Higher scores indicate worse outcome. Minimum score = 0; maximum score = 49. Higher scores indicate worse outcome.
Generalised Anxiety Disorder assessment 7-items | assessed at 3, 6, 9 and 12-month follow-up
  A brief self-reported measure of generalised anxiety symptoms using 4-point Likert scales based on diagnostic criteria. Minimum score = 0; maximum score = 21. Higher scores indicate worse outcome.
Patient Health Questionnaire 9-items | assessed at 3, 6, 9 and 12-month follow-up
  Assesses symptoms of depression using self-reported 4-point Likert scales based on diagnostic criteria for major depression. Minimum score = 0; maximum score = 27. Higher scores indicate worse outcome.
Euroqol 5-dimensions 3-levels | assessed at 3, 6, 9 and 12-month follow-up
  a self-reported assessment of five key dimensions of health-related quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The youth version will be used for participants under 16 years old. Minimum score = 0; maximum score = 1. Higher scores indicate better outcome.
Patient-Reported Outcomes Measurement Information System, Satisfaction with Social Roles and Activities | assessed at 3, 6, 9 and 12-month follow-up
  Assesses satisfaction with performing one's usual social roles and activities. It, therefore, acts as a measure of social engagement which can be heavily impacted by brain tumour diagnosis and treatment. Minimum score = 8; maximum score = 40. Higher scores indicate worse outcome.
Strengths and Difficulties Questionnaire 25-item | assessed at 3, 6, 9 and 12-month follow-up
  A patient and parent/carer-completed brief measure of behavioural and emotional functioning. Minimum score = 0; maximum score = 50. Higher scores indicate better outcome.
Client Service Receipt Inventory | assessed at 3, 6, 9 and 12-month follow-up
  A research instrument developed to collect information on service receipt, service-related issues and income. In addition, the Client Service Receipt Inventory collects information on school attendance in the 3-months prior to assessment.
Experiential interviews | assessed at 3- and 6-month follow-up
  Participant experiences of treatment as described in semi-structured qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Thomas, DClinPsy, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Sophie Thomas, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participant consent will be requested for the publication of anonymised questionnaire data onto the Figshare research repository, in line with current research transparency best practice guidance (Miguel et al., 2014; Nosek et al., 2015).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be published after the trial results are published.
Access Criteria: Data will be openly available from Figshare

REFERENCES:
- [Derived] Malins S, Owen R, Wright I, Borrill H, Limond J, Gibson F, Grundy RG, Bailey S, Clifford SC, Lowis S, Lemon J, Hayes L, Thomas S. Acceptance and commitment therapy for young brain tumour survivors: study protocol for an acceptability and feasibility trial. BMJ Open. 2021 Jun 1;11(6):e051091. doi: 10.1136/bmjopen-2021-051091. PMID 34078638